CLINICAL TRIAL: NCT02971332
Title: STARR With Contour Transtar for Obstructed Defecation Syndrome: Long Term Results
Brief Title: Long Term Results of STARR With Contour Transtar
Acronym: LTSTARR
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, MD, PhD, FACS, MD, PhD, FACS, University of Roma La Sapienza
Other Study IDs: STR016a
Record Dates: First submitted 2016-11-20; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Rectal Prolapse; Rectocele; Intussusception of Rectum
MeSH Terms: conditions — Rectal Prolapse; Rectocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: Patients candidated to STARR after the failure of medical and dietary therapy and after a complete radiological and functional study.
  Interventions: Procedure: Stapled Transanal Rectal Resection

INTERVENTIONS:
Procedure: Stapled Transanal Rectal Resection — The prolapsed tissue is pulled out through the CAD using e gauze pad and Allis forceps; this allows us to identify the extent of the prolapse to be resected. Four to five parachute stitches are then apposed circumferentially, like parachute cords, at the apex of the prolapse, in order to control the tissue during resection. The prolapse is then opened longitudinally at 3 o'clock with the electric scalpel between two Kocher clamps. Two traction stitches are applied at the deep vertex of the prolapse, one for each Kocher apex.
  The longitudinal opening then allows the surgeon to begin circumferential resection of the rectum by pulling on the parachute stitches. This maneuver is performed counterclockwise using an average of 4-6 recharges, with care to always place the stapler at the base of the prolapse. The resected specimen was always inspected before the end of the procedure.
  Other Names: STARR

SUMMARY:
Obstructed defecation syndrome (ODS) is a widespread and disabling syndrome. With this study the investigators want to evaluate the long term results of Stapled Transanal Rectal Resection (STARR) performed with Contour Transtar device in the treatment of ODS. A re-evaluation of 113 patients subjected to STARR from June 2007 to January 2010 was conducted.

ELIGIBILITY:
Inclusion Criteria:

* ODS
* presence of a rectocele that did not empty and/or a recto-rectal or recto-anal intussusception.

Exclusion Criteria:

* anal sphincter contractile deficiency
* previous rectal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic ODS after failure of medical and dietary therapy and with the presence determined through cinedefecography of a rectocele that did not empty and/or a recto-rectal or recto-anal intussusception, in the absence of anal sphincter contractile deficiency
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
degree of constipation | 6 months
  Cleveland Clinic Constipation Score
degree of constipation | 5 years
  Cleveland Clinic Constipation Score

SECONDARY OUTCOMES:
Surgical Complications | 0-6 months
  intraoperative and postoperative surgical complications

OTHER OUTCOMES:
Defecatory aids | 6 months
  the use of laxatives or digitation to defecate
Defecatory aids | 5 years
  the use of laxatives or digitation to defecate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mari FS, Pezzatini M, Gasparrini M, Antonio B. STARR with Contour Transtar for Obstructed Defecation Syndrome: Long-Term Results. World J Surg. 2017 Nov;41(11):2906-2911. doi: 10.1007/s00268-017-4084-6. PMID 28600694